CLINICAL TRIAL: NCT05234125
Title: A Randomized Control Trial to Improve Metabolic Outcomes in African American Pregnant Women
Brief Title: Better Lifestyle Counseling for African American Women During Pregnancy
Acronym: BETTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Office of Research on Women's Health (ORWH) (NIH); Office of Behavioral and Social Sciences Research (OBSSR) (NIH)
Responsible Party: Principal Investigator, Bilgay Izci Balserak, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-0918; R01MD015724 (NIH)
Record Dates: First submitted 2022-01-15; First posted 2022-02-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Overweight or Obesity; Pregnancy Related; Sleep Disturbances; Sleep Hygiene; Pregnancy Complications; Diversity; Stress, Psychological; Fitness Trackers; Exercise; African Americans; Disparities in Pregnancy Complications; Sleep Disparities
Keywords: Sleep, Pregnancy, Intervention, glucose metabolism,
MeSH Terms: conditions — Overweight; Obesity; Parasomnias; Sleep Hygiene; Pregnancy Complications; Stress, Psychological; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Sleep hygiene practices and cognitive-behavioral principles
  Interventions: Behavioral: Better
- Attention control (Placebo Comparator): Training about pregnancy issues
  Interventions: Behavioral: Birth Prep

INTERVENTIONS:
Behavioral: Better — It is a nonpharmacologic sleep intervention to improve maternal glucose metabolism in African American Pregnant Women (AAPW). Sleep BETTER is composed of sleep hygiene practices and cognitive-behavioral principles.
  Other Names: Sleep BETTER
  Arms: Intervention arm
Behavioral: Birth Prep — The intervention involves training about pregnancy-related issues, and follow up
  Arms: Attention control

SUMMARY:
The purpose of this randomized controlled trial is to establish the effectiveness of a culturally targeted and individually tailored behavioral intervention to promote maternal glucose metabolism in African American women.

DETAILED DESCRIPTION:
This is a randomized controlled parallel-group trial with two arms. Potential subjects will be identified from the OB Clinics at UI health systems, the University of Illinois at Chicago. After baseline assessments, the subjects will be randomized to the attention control arm (Birth-Prep) or BETTER intervention.

ELIGIBILITY:
Inclusion Criteria:

* African American pregnant woman.
* Women between 16 and 22 GWs.
* Overweight or obese - pregravid Body Mass Index >25.0 kg/m2.
* Singleton gestation.
* Established prenatal care at The University of Illinois Hospital & Health Sciences.
* System Obstetric (UIHHSS' OB) clinics. Able to understand, speak and write in English.

Exclusion Criteria:

* Multiple gestations.
* Night-shift work.
* Diagnosed sleep disorders.
* Known fetal chromosomal or anatomical abnormalities.
* Diagnosed mood disorders.
* Gestational diabetes in early pregnancy.
* Glycated Hemoglobin (HbA1c) ≥ 6.5%.
* Hypoglycemic medications.
* Stimulant medication or taking a sleeping aid.
* Active drug abuse/excessive alcohol intake.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Fasting Glucose at baseline | 16-22 Gestational Weeks (GWs)
  A fasting blood sample for glucose will be collected
Fasting Glucose | 28-32 Gestational Weeks (GWs)
  A fasting blood sample for glucose will be collected

SECONDARY OUTCOMES:
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at baseline | 16-22 Gestational Weeks
  Insulin Resistance
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 28-32 Gestational Weeks
  Insulin Resistance
Glucose Area Under the Curve at baseline | 16-22 Gestational Weeks
  Glucose tolerance
Glucose Area Under the Curve | 28-32 Gestational Weeks
  Glucose tolerance
Glucose Area Under the Curve | 34-36 Gestational Weeks
  Glucose tolerance
Sleep Quality - Self-reported of sleep quality at the baseline "before the intervention" | 16-22 Gestational Weeks
  Self-reported sleep quality over the past month will be assessed by using Pittsburgh Sleep Quality Index (PSQI) Questionnaire.
  * It is a 19 self-rated questions, 4-point Likert-scale. Each score ranges from 0 - 3.
  * It is a self-report measure that assesses sleep quality and severity of specific sleep related complaints over the previous month.
  * Higher score=poorer sleep quality.
Sleep Quality - Self-reported of sleep quality | 28-32 Gestational Weeks
  Self-reported sleep quality over the past month will be assessed by using Pittsburgh Sleep Quality Index (PSQI) Questionnaire.
  * It is a 19 self-rated questions, 4-point Likert-scale. Each score ranges from 0 - 3.
  * It is a self-report measure that assesses sleep quality and severity of specific sleep related complaints over the previous month.
  * Higher score=poorer sleep quality.
Sleep Quality - Self-reported of sleep quality | 34-36 Gestational Weeks
  Self-reported sleep quality over the past month will be assessed by using Pittsburgh Sleep Quality Index (PSQI) Questionnaire.
  * It is a 19 self-rated questions, 4-point Likert-scale. Each score ranges from 0 - 3.
  * It is a self-report measure that assesses sleep quality and severity of specific sleep related complaints over the previous month.
  * Higher score=poorer sleep quality.
Sleep duration and sleep timing - Subjectively and Objectively Assessment at the baseline "before the intervention" | 16-22 Gestational Weeks
  sleep duration will be assessed using a wearable device (Fitbit Charge 4) accompanied by a sleep diary.
  Sleep timing (midpoint) will be calculated as the halfway point between bedtime and rise time.
Sleep duration and sleep timing - Subjective and Objective Assessment | 28-32 Gestational Weeks
  sleep duration will be assessed using a wearable device (Fitbit Charge 4) accompanied by a sleep diary.
  Sleep timing (midpoint) will be calculated as the halfway point between bedtime and rise time.
Sleep duration and sleep timing - Subjective and Objective Assessment | 34-36 Gestational Weeks
  Sleep duration will be assessed using a wearable device (Fitbit Charge 4) accompanied by a sleep diary. Sleep timing (midpoint) will be calculated as the halfway point between bedtime and rise time.
Medical Records Extraction Form | "post delivery, up to 3 months post intervention"
  Maternal-fetal outcomes will be assesses by reviewing participants' medical records and report the incidence of: newborn's hypoglycemia, macrosomia, & intensive care admission - preterm and cesarean deliveries, preeclampsia, gestational hypertension and any other important events.
  In addition, Apgar scores and birth weight will be reported.
  Pregnancy outcomes will be obtained from medical charts to understand if there are differences regarding these outcomes between the BETTER and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bilgay Izci Balserak, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Irsheed GA, Steffen A, Quinn L, Chen P, Maharana S, Burke L, Borbas L, Alameda G, Maganuru R, Balserak BI. Poor Sleep Environment and Increased Insulin Resistance in Black/African American Pregnant Women: A Cross-Sectional Study. J Racial Ethn Health Disparities. 2025 Nov 18. doi: 10.1007/s40615-025-02747-5. Online ahead of print. PMID 41254328